CLINICAL TRIAL: NCT03881150
Title: Effectiveness of a Hybrid Cardiac Rehabilitation Program for Coronary Artery Disease Patients. Randomized, Multicenter, Non-inferiority Clinical Trial in a Low-resource Setting. HYCARET Study
Brief Title: Hybrid Cardiac Rehabilitation Trial
Acronym: HYCARET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Pamela Serón, Professor, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fondecyt 1181734
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Cardiac rehabilitation; Exercise; Coronary Artery Disease; Mobile technology
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Motor Activity | interventions — Counseling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Cardiac Rehabilitation (Experimental): This intervention is adapted from the "Cardiac Rehabilitation Delivery Model for Low-Resource Settings" proposed by the International Council of Cardiovascular Prevention and Rehabilitation Consensus Statement. This program will be delivered by an exercise specialist (physiotherapist) and the principal purposes of the exercise sessions is to develop patient self-management related to the physical activity habit, and educate them how to monitor exercise intensity at home and in daily life. The program include 10 face-to-face exercise sessions and a transition to unsupervised phase using mobile technology.
  Counseling is considered about physical activity, diet, smoking, and medication compliance.
  Interventions: Other: Comprehensive assessment; Other: Counseling; Other: Exercise sessions in hybrid program; Other: Transition to unsupervised phase
- Standard Cardiac Rehabilitation (Active Comparator): The participants in the control group will receive the standard cardiac rehabilitation that is delivered in participating centers. These programs accounts with physicians, nurses, nutritionists and physiotherapists. The programs will be standardized in participating centers in accordance with currents guidelines (only 18-22 face-to-face exercise sessions). Differentially, this programs provide, group education sessions about physical activity, diet, smoking, and medication compliance (without counseling).
  Interventions: Other: Comprehensive assessment; Other: Group education; Other: Exercise sessions in standard program

INTERVENTIONS:
Other: Comprehensive assessment — Includes evaluation about physical activity, diet, tobacco consumption, overweight/obesity, blood pressure, self-efficacy, and medications. Additionally, levels of lipids and glycaemia will be reviewed from clinical chart.
Other: Counseling — Physical activity, diet, smoking, and medication compliance counseling will be provided by the physiotherapist across exercise sessions, using a self-efficacy approach. A booklet was designed in order to support the individual counseling.
  Arms: Hybrid Cardiac Rehabilitation
Other: Group education — Group education sessions about physical activity, diet, smoking, and medication compliance (without individual counseling), as actually performed in each center.
  Arms: Standard Cardiac Rehabilitation
Other: Exercise sessions in hybrid program — 10 supervised exercise sessions over 4-6 weeks of aerobic and resistance training will ensue, supervised by a physiotherapist. Exercise sessions are 10 minutes in duration at the beginning of the program, and are progressed to 60 minutes by the end as tolerated.
  Intensity of exercise will be moderate.
  Arms: Hybrid Cardiac Rehabilitation
Other: Exercise sessions in standard program — 18-22 supervised exercise sessions are delivered over the 8-12 week program. These sessions include aerobic and resistance training and a similar progression of duration as the experimental group.
  Intensity of exercise will be moderate.
  Arms: Standard Cardiac Rehabilitation
Other: Transition to unsupervised phase — After 4-6 weeks with face-to-face exercise sessions in hybrid program, all patients will be monitored through mobile technology. Delivery methods will include voice calls biweekly, and text messaging three per week through to 10-12 weeks from program initiation. The content will promote physical activity, healthy diet, and medication adherence.
  Arms: Hybrid Cardiac Rehabilitation

SUMMARY:
This clinical trial aim to evaluate if the prevention of recurrent cardiovascular events is not inferior in the hybrid mobile and exercise-based cardiac rehabilitation programs in comparison to the standard cardiac rehabilitation program.

DETAILED DESCRIPTION:
Background: Cardiac rehabilitation (CR) programs are well established, as their effectiveness and cost-effectiveness is proven. In spite of this, CR remains under-utilized, especially in middle and low-resource settings such as Latin America. As the highest rates of mortality and disability-adjusted life-years in the world are caused by cardiovascular diseases, with a corresponding major impact on economies, there is an urgent need to create more accessible CR delivery models to reach all patients in need. This trial aims to evaluate if the prevention of recurrent cardiovascular events is not inferior in a hybrid cardiac rehabilitation program compared to a standard program.

Method and analysis: A non-inferiority, pragmatic, multicenter, parallel (1:1), single blinded, randomized clinical trial will be conducted. 314 patients with coronary artery disease will be recruited consecutively. Participants will be randomized to hybrid or standard rehabilitation programs. The hybrid CR program includes 10 supervised exercise sessions and individualized lifestyle counseling by a physiotherapist, with a transition after 4-6 weeks to unsupervised delivery via text messages and phone calls. The standard CR consists of 18-22 supervised exercise sessions, as well as group education sessions about lifestyle. The intervention in both groups will be by 12 weeks. The primary outcome is a composite of cardiovascular mortality and hospitalizations due to cardiovascular causes. Secondary outcomes are cardiovascular risk factor control, exercise capacity, adherence to physical activity and diet recommendations, health-related quality of life and exercise-related adverse events. The outcomes will be measured at the end of intervention, at 6 months, and at 12-month follow-up from recruitment. The primary outcome will be tracked through the end of the trial. The sample size was calculated considering 5% of the non-inferiority limit. Per protocol and intention-to-treat analysis will be undertaken. A survival analysis will be run for the primary outcome.

Ethics and dissemination: The corresponding ethical committees at the sponsor institution and each center where participants will be recruited approved the study protocol and the Informed Consent form. Research findings will be published in peer-reviewed journals. Additionally, scientific results will be disseminated among stakeholders and national policy-makers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year old or over.
* Patient with coronary artery disease, including Acute Coronary Syndrome (Unstable Angina, Myocardial infarction with or without ST elevation) or stable coronary vessel disease diagnosed by angiography or a stress test.
* Patient treated medically (i.e., medication only) or by thrombolysis, angioplasty, or revascularization surgery.
* Patient with physician referral, that can start CR between 2 weeks and 2 months from their event, diagnosis or procedure.
* Patient able to attend the health center almost twice a week over three months.
* Patient owns a mobile phone.
* Patient that consents to participate in the study through signing an informed consent form.

Exclusion Criteria:

* Patient has a planned repeat cardiac or other procedure in next 12 months.
* Explicit contraindication to perform exercise based on American College of Sport Medicine.
* Patients with comorbidities that would interfere with ability to engage in cardiac rehabilitation such as dementia, blindness, deafness, serious mental illness, or frailty.
* Musculoskeletal disease that precludes the patient from performing exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Recurrent cardiovascular events | 12 months (or more for first recruited participants, but until 36 months).
  Composite of cardiovascular mortality (defined as death by stroke, myocardial infarction or heart failure) and hospitalizations due to a cardiovascular cause (non-fatal stroke, non-fatal myocardial infarction, heart failure, and need for revascularization surgery)

SECONDARY OUTCOMES:
Health-related quality of life | Baseline, end of intervention (8-12 weeks), 6 months, and 12 months.
  HeartQoL as disease-specific and EuroQol five-dimensional three-level (EQ-5D-3L) as generic instrument will be administered
Functional exercise capacity | Baseline, end of intervention (8-12 weeks), 6 months, and 12 months
  In meters (mts) obtained in the 6 Minute Walking Test
Grip strength | Baseline, end of intervention (8-12 weeks), 6 months, and 12 months
  In kilograms (kgs) obtained by dynamometry
Adherence to physical activity recommendations | Baseline, end of intervention (8-12 weeks), 6 months, and 12 months.
  The International Physical Activity Questionnaire (IPAQ) will be administered. This instrument can quantify the energy spent in MET-minutes/week for categorization in accordance with the World Health Organization recommendation: An adults 18 years old or over adheres when perform 150 minutes of moderate-intensity aerobic activity or 75 minutes of vigorous activity per week, or a combination of both.
Adherence to diet recommendations | Baseline, end of intervention (8-12 weeks), 6 months, and 12 months.
  Trained personnel will administer the Mediterranean Dietary Index for Chilean population (Chile-MDI). Participants recall the frequency of consumption of 14 food groups. This instrument had been validated. Scores range from 0 to 14 points, indicating absence and maximum adherence, respectively.
Return-to-work | End of intervention (8-12 weeks), 6 months, and 12 months
  Concordance between desired and actual work status at assessment
Body Mass Index (BMI) | Baseline, end of intervention (8-12 weeks), 6 months, and 12 months
  Weight and height will be combined to report BMI in kg/m2
Waist circumference | Baseline, end of intervention (8-12 weeks), 6 months, and 12 months
  In centimeters (cms)
Blood Pressure | Baseline, end of intervention (8-12 weeks), 6 months, and 12 months
  In millimeters of mercury (mmHg)
Adherence | End of intervention (8-12 weeks)
  Percentage of attendance at supervised sessions planned. Also adherence to the calls in the intervention group will be collect.
Exercise related adverse events | End of intervention (8-12 weeks)
  Counting adverse events during exercise, such as myocardial ischemia or malignant arrhythmias, will be registered. Serious adverse event, as death in the exercise session, will be registered and reported to corresponding ethic committee and monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Seron, PhD, Principal Investigator — Universidad de La Frontera
Locations (6):
- Chile (6):
  - Universidad de La Frontera, Temuco, Región de la Araucanía
  - Hospital Regional de Antofagasta, Antofagasta
  - Complejo Hospitalario San José, Santiago
  - Hospital Clínico Universidad de Chile, Santiago
  - Hospital San Borja Arriarán, Santiago
  - Hospital San Juan de Dios, Santiago

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the main results article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 6 months following main results article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For individual participant data meta-analysis. Proposals should be directed to Principal Investigator. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Seron P, Oliveros MJ, Marzuca-Nassr GN, Morales G, Roman C, Munoz SR, Galvez M, Latin G, Marileo T, Molina JP, Navarro R, Sepulveda P, Lanas F, Saavedra N, Ulloa C, Grace SL; HYCARET Investigators. Hybrid Cardiac Rehabilitation Program in a Low-Resource Setting: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2350301. doi: 10.1001/jamanetworkopen.2023.50301. PMID 38194236
- [Derived] Seron P, Oliveros MJ, Marzuca-Nassr GN, Lanas F, Morales G, Roman C, Munoz SR, Saavedra N, Grace SL. Hybrid cardiac rehabilitation trial (HYCARET): protocol of a randomised, multicentre, non-inferiority trial in South America. BMJ Open. 2019 Oct 28;9(10):e031213. doi: 10.1136/bmjopen-2019-031213. PMID 31662385